CLINICAL TRIAL: NCT06280040
Title: Longitudinal Follow-Up of Retinopathy and Opticopathy After Treatment With Hypofractionated Stereotactic Photon Radiotherapy Due to Uveal Melanoma
Brief Title: Longitudinal Follow-Up of Patients Treated With Hypofractionated Stereotactic Photon Radiotherapy Due to Uveal Melanoma
Status: Recruiting | Type: Observational
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Reinhard Told, MD, PHD, Medical University of Vienna
Other Study IDs: UM Longitudinal 1942/2022
Record Dates: First submitted 2024-02-20; First posted 2024-02-28 (Actual); Last update posted 2024-03-06 (Actual); Status verified 2024-03

CONDITIONS: Uveal Melanoma
MeSH Terms: conditions — Uveal Melanoma | interventions — Physical Examination

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Uveal Melanoma: Patients with newly diagnosed uveal melanoma, which will be treated with hypofractionated stereotactic photon radiotherapy as clinical routine.
  Interventions: Diagnostic Test: Clinical examination and multimodal ocular imaging

INTERVENTIONS:
Diagnostic Test: Clinical examination and multimodal ocular imaging — Imaging consists of sonography, fundus photography, oximeter, optical coherence tomography angiography, and Microperimetry.

SUMMARY:
The purpose of this study is to evaluate the incidence and severity of retinopathy and opticopathy one year after treatment with hypofractionated stereotactic photon radiotherapy due to uveal melanoma. Patients will be imaged before radiation, as well as 3, 6, 9 and 12 months after radiation using sonography funds photography, optical coherence tomography angiography, oximeter and microperimetry.

ELIGIBILITY:
Inclusion Criteria:

* Patients with newly diagnosed uveal melanoma, who will be treated with hypofractionated stereotactic photon radiotherapy as part of clinical routine.

Exclusion Criteria:

* unwillingness to participate in the study
* severe media opacity

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with newly diagnosed uveal melanoma, who will be treated with hypofractionated stereotactic photon radiotherapy as part of clinical routine, will be included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2023-11-23 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Incidence and Severity of Retinopathy | 1 year
  Incidence and severity of retinopathy will be evaluated as non-perfusion areas on optical coherence tomography angiography

SECONDARY OUTCOMES:
Incidence and Severity of Opticopathy | 1 year
  Incidence and severity of retinopathy will be evaluated on clinical examination and fundus photography
Functional Outcome | 1 year
  Functional outcome will be evaluated as mean retinal sensitivity.
Incidence and Severity of Retinopathy and Opticopathy in oximeter | 1 year
  Incidence and severity of retinopathy and opticopathy will be evaluated using oxygen saturation

CONTACTS AND LOCATIONS:
Overall Officials: Reinhard Told, MD, PhD, Principal Investigator — Department for Ophthalmology and Optometry, Medical University of Vienna
Locations (1):
- Department of Ophthalmology and Optometry, Medical University Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: Undecided